CLINICAL TRIAL: NCT00375154
Title: Noninvasive Positive-pressure Ventilation (NPPV) for Acute Respiratory Failure in Out-of-hospital Patients: a Multicenter, Prospective, Randomized Controlled Trial
Brief Title: HERMES STUDY: Study on the Feasibility and Efficiency of Noninvasive Positive-Pressure Ventilation (NPPV) in Prehospital Care
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: major difficulties in training investigators in other centers
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Collaborators: Frederic Thys,MD,PhD (Unknown)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: URGPROT1
Record Dates: First submitted 2006-09-11; First posted 2006-09-12 (Estimated); Last update posted 2011-07-20 (Estimated); Status verified 2011-07

CONDITIONS: ARF Secondary to COPD Exacerbation; ARF Secondary to Cardiogenic Acute Pulmonary Oedema
Keywords: Acute respiratory failure; Prehospital care; Noninvasive ventilation; Emergency
MeSH Terms: conditions — Emergencies

INTERVENTIONS:
Device: Noninvasive Positive-Pressure Ventilation (NPPV)

SUMMARY:
The purpose of this study is determine if NPPV can be performed in a pre-hospital setting very early after onset of dyspnea with a similar benefit in need of intubation and mortality as in previous study in hospital context and if early NPPV intervention have a real, rather standard medical therapy, value, both on objectively measured parameters and on patient's clinical status.

DETAILED DESCRIPTION:
Noninvasive positive-pressure ventilation (NPPV) is increasingly being used in the care of patients suffering acute respiratory failure. High-level evidence supports the use of NPPV in this setting. With selected patients, NPPV decreases the rate of intubation, mortality and nosocomial infections. NPPV obviates intubation in > 50 % of appropriately selected patients. Both nasal and oronasal interfaces have been successfully used to apply NPPV, but the oronasal (or facial) interface is often used for acute respiratory failure. Any ventilator and ventilator mode can be used to apply NPPV, but in practice, portable pressure ventilators and pressure-support mode are most commonly used.

In acute setting, this therapy must be applied as soon as possible after the onset of problem. With our research team, we have demonstrated that NPPV can be used with success in an emergency department. In our experience, when NPPV was early used, part of the patients improved rapidly and was could be admitted to a general ward. An interesting fact is that the time to improve clinical situation is short and we can postulated than NPPV application in emergency department may be used as a "clinical triage". We have also demonstrated that early application of bi-level NPPV to patients with acute respiratory failure due to acute exacerbation of COPD or APO leads to a rapid improvement in clinical status and blood gases that differs substantially from the evolution of similar patients treated with conventional medical therapy and a placebo NPPV device.

Currently, we have very few data on the real utility to use of NPPV in Out-of-Hospital patients with acute respiratory failure managed by medical team of pre-hospital care despite the fact that this approach decreased the delay of application of a efficient ventilator support. A prior study of Craven and coll. has demonstrated that NPPV helps relieve dyspnea in patients with suspected congestive heart failure.

We can postulate that a shorter delay between onset of symptomatology and application of NPPV increased the part of selected patient with good clinical outcome (intubation, need of intensive care).

Comparisons :

Patients with COPD, APO with standard medical therapy + NPPV compared to patients with standard medical therapy alone in pre-hospital setting.

ELIGIBILITY:
Inclusion Criteria:

* Out-of-hospital patients with acute respiratory failure
* only patients with COPD, APO are included.
* Patients are eligible into the study if the attending physician judged that the need of a mechanical ventilatory support is imminent.
* Patients not improving under usual treatment

Exclusion Criteria:

* An immediate indication for endotracheal intubation (respiratory and/or cardiac arrest).
* Major unrest.
* Hemodynamic instability despite a fluid challenge (500 ml of colloids).
* Facial or thoracic trauma.
* Lack of cooperation.
* Difficult adaptation of facial mask to patient's facial anatomy.
* Clinical suspicion of pulmonary embolism.
* Retrosternal pain suggestive of a myocardial ischemia
* If the investigators are not available.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2006-08

PRIMARY OUTCOMES:
Difference in the number of in each arm of the study failing at the time of admission in emergency department.

SECONDARY OUTCOMES:
Effects of the ventilatory mode on the clinical and arterial-blood gas parameters
Hospital mortality
Admission to the ICU, the length of ED stay, the length of ICU stay and the length of hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Frederic C Thys, MD,PhD, Study Chair — Emergency Department; Cliniques Universitaires Saint-Luc; Université Catholique de Louvain
Locations (8):
- Belgium (8):
  - Emergency Department; Cliniques Universitaires Saint-Luc, Brussels
  - CHU Brugman-Schaerbeek, Brussels
  - Hôpital de Dinant, Dinant
  - Cliniques Notre Dame de Gosselies, Gosselies
  - Citadelle CHR Liège, Liège
  - CHR Namur, Namur
  - CHR de Tournai, Tournai
  - Cliniques Universitaires de Mont-Godinne ; Université Catholique de Louvain, Yvoir

REFERENCES:
- [Background] Thys F, Roeseler J, Reynaert M, Liistro G, Rodenstein DO. Noninvasive ventilation for acute respiratory failure: a prospective randomised placebo-controlled trial. Eur Respir J. 2002 Sep;20(3):545-55. doi: 10.1183/09031936.02.00287402. PMID 12358327
- [Background] Thys F, Roeseler J, Delaere S, Palavecino L, El Gariani A, Marion E, Meert P, Danse E, D'Hoore W, Reynaert M. Two-level non-invasive positive pressure ventilation in the initial treatment of acute respiratory failure in an emergency department. Eur J Emerg Med. 1999 Sep;6(3):207-14. PMID 10622384
- [Background] Vanpee D, Delaunois L, Lheureux P, Thys F, Sabbe M, Meulemans A, Stroobants J, Dorio V, Gillet JB. Survey of non-invasive ventilation for acute exacerbation of chronic obstructive pulmonary disease patients in emergency departments in Belgium. Eur J Emerg Med. 2002 Sep;9(3):217-24. doi: 10.1097/00063110-200209000-00003. PMID 12394617
- [Background] Craven RA, Singletary N, Bosken L, Sewell E, Payne M, Lipsey R. Use of bilevel positive airway pressure in out-of-hospital patients. Acad Emerg Med. 2000 Sep;7(9):1065-8. doi: 10.1111/j.1553-2712.2000.tb02102.x. PMID 11044006